CLINICAL TRIAL: NCT03924882
Title: A Phase II Study of Anlotinib for Patients With Platinum Resistant or Refractory Ovarian Cancer
Brief Title: Anlotinib for Patients With Platinum Resistant or Refractory Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOC
Record Dates: First submitted 2019-04-21; First posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Ovarian Cancer
Keywords: Anlotinib; Ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Anlotinib — Anlotinib QD po and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent

SUMMARY:
The purpose of the study is to evaluate the efficacy and toxicity of anlotinib in patients with platinum resistant or refractory ovarian cancer

DETAILED DESCRIPTION:
Ovarian cancer is the leading cause of death for patients with gynecologic malignancies. In most cases, the disease is diagnosed at an advanced stage and approximately 75% of patients will eventually experience disease recurrence. However, the overall response rates of second-line chemotherapy for recurrent ovarian cancer are only 20-27%. Therefore, it is important to seek alternative agent that can improve the outcome. Anlotinib is a new, orally administered tyrosine kinase inhibitor that targets VEGFR,FGFR,PDGFR,and c-kit,. The preclinical studies suggest anlotinib may be effective in other cancers such as ovarian cancer. Therefore, the purpose of this study is to test the efficacy and safety of the study drug anlotinib.

ELIGIBILITY:
Inclusion Criteria:

1. Female, age ≥18 years and ≤70 years, signed informed consent.
2. Histologically or pathologically confirmed diagnosis of epithelial carcinoma of the ovary.
3. Platinum resistant ovarian cancer (defined as relapsing within 6 months after the last administration of platinum-based chemotherapy) OR platinum refractory ovarian cancer (defined as progressing while on a platinum-based chemotherapy)
4. At least treated with one line of platinum-based chemotherapy
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
6. Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 version or CA125
7. Patients must have a life expectancy of at least 3 months.
8. Patients must have adequate organ function.

Exclusion Criteria:

1. Had prior exposure to anlotinib or has known allegies to any of the excipients, Inadequately controlled hypertension
2. History of myocardial infarction, or unstable angina, or New York Heart Association (NYHA) Grade III-IV within 6 months prior to Day 1.
3. History of abdominal fistula or gastrointestinal perforation within 28 days prior to Day 1
4. Major surgical procedure within 28 days prior to Day 1, Serious, non-healing wound, active ulcer, bowel obstruction within 28 days prior to Day 1
5. Symptomatic central nervous system (CNS) metastasis

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-04-25 (Estimated); Primary Completion 2021-04-25 (Estimated); Study Completion 2022-04-25 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to three years
  Objective response rate defined as confirmed complete response or partial response under RECIST 1.1 criteria. CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. To be assigned a status of CR or PR, changes in tumor measurements must be confirmed by repeat assessments performed no fewer than 4 weeks after the response criteria are first met.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to three years
Duration of Response | Up to three years
Frequency and severity of adverse effects as defined by CTCAE version 4.03 | 30 days after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Jianwei Zhou, M.D., Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China